CLINICAL TRIAL: NCT00411437
Title: A Randomized, Double-Blind, Placebo-Controlled, Three Arm Study To Evaluate The Effects Of Tolterodine ER 4 mg Vs. Placebo Vs. Oxybutynin ER On Memory And Other Cognitive Abilities In Elderly Subjects
Brief Title: Effects Of Detrol LA On Memory And Cognition In Elderly Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6121154
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Memory; Cognition
MeSH Terms: interventions — Tolterodine Tartrate

INTERVENTIONS:
Drug: Tolterodine ER
Drug: Oxybutynin ER

SUMMARY:
The primary purpose of the trial is to show that tolterodine ER has no effect on memory and other cognitive abilities in an elderly population

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with age of 65 - 75 years
* Having a score of greater than or equal to 26 on the Mini-Mental State Exam (MMSE)

Exclusion Criteria:

* Current or history of bladder outlet obstruction. Previous history of acute urinary retention requiring catheterization, or severe voiding difficulties in the judgment of the investigator, prior to randomization
* Significant hepatic or renal disease, defined as twice the upper limit of the reference ranges regarding serum concentrations of AST, ALT, ALP, urea nitrogen, or creatinine

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 220
Dates: Start 2006-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Delayed Recall on the Name-Face Association Test at Week 3 (tolterodine ER vs. placebo) - Number of correct responses to the test

SECONDARY OUTCOMES:
1. Cognitive effects of tolterodine ER vs. placebo at Weeks 1 and 2 on Delayed Recall on the Name-Face Association Test - Number of correct responses to the
test 2. Cognitive effects of tolterodine ER vs. oxybutynin ER and oxybutynin ER vs. placebo at Weeks 1, 2, and 3 on Delayed Recall on the Name-Face
Association Test - Number of correct responses to the test 3. Other cognitive effects in the following three paired comparisons: tolterodine ER vs. placebo;
tolterodine ER vs. oxybutynin ER; and oxybutynin ER vs. placebo on: 3a) Delayed Recall Domain (Verbal and Visual) at Weeks 1, 2, and 3: 3a_i) Delayed Recall on
the First-Last Name Association Test - Number of correct responses to the test 3a_ii) Misplaced Objects Test - Number of correct recalls at the first attempt 3b)
Immediate Recall Domain at Weeks 1, 2, and 3: 3b_i) Immediate Recall on the Name-Face Association Test - Number of correct responses to the test in the first
acquisition - Number of correct responses to the test in the second acquisition 3b_ii) Immediate Recall on the First-Last Name Association Test - Number of
correct responses to the test in the first acquisition - Number of correct responses to the test in the second acquisition 3b_iii) Facial Recognition Test - Number of
correct responses before first miss - Total correct responses 3c) Visual Attention and Memory Domain at Weeks 1, 2, and 3: 3c_i) Matching-to-Sample Test -
Throughput (number of correct responses / minute) 3c_ii) Visual Sequence Comparison Test - Throughput (number of correct responses / minute) 3d)
Psychomotor/Reaction-Time Domain at Weeks 1, 2, and 3: 3d_i) Divided Attention Test (response speed to visual monitoring task alone) - Median response time for
correct responses (seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121154&StudyName=Effects%20Of%20Detrol%20LA%20On%20Memory%20And%20Cognition%20In%20Elderly%20Population